CLINICAL TRIAL: NCT04701736
Title: A Randomized Controlled Trial to Assess the Influence of a Picture-Based Antiemetic Medication Calendar on Medication-Taking Behavior in Adults Receiving Chemotherapy
Brief Title: A Trial to Assess the Influence of a Pictorial Medication Calendar on Medication Taking Behaviour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Waterloo (Other); Medbuy Corporation (Unknown); London Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 107084
Record Dates: First submitted 2017-08-25; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2019-12

CONDITIONS: Cancer; Chemotherapy; Medication Adherence
Keywords: patient adherence; chemotherapy; pictorial aid; complex medication regimen; cancer
MeSH Terms: conditions — Neoplasms; Medication Adherence; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care (No Intervention): Routine care consists of an oncology pharmacist counselling the patient on supportive care medications prior to the patient getting his or her prescription dispensed.
- Intervention (Active Comparator): The intervention group will encompass the oncology pharmacist using the computer system to print a Picture Medication Calendar for the patient and use the calendar to explain supportive medications, in addition to routine care.
  Interventions: Device: Picture Medication Calendar

INTERVENTIONS:
Device: Picture Medication Calendar
  Arms: Intervention

SUMMARY:
Determine if an oncology pictorial medication calendar will improve patient adherence to oncology supportive care medication regimens for adult patients receiving adjuvant or neo-adjuvant chemotherapy treatment for cancer.

DETAILED DESCRIPTION:
Primary Objective: In order to evaluate the impact of such an approach on adherence, a prospective, open-label, randomized controlled pilot trial (RCT) was carried out to determine if a picture-based medication calendar would improve patient adherence to antiemetic medication regimens for adult patients receiving chemotherapy treatment for solid organ tumor origins.

The secondary objectives were: 1) to assess medication use and self-efficacy parameters, 2) to determine patient comfort with antiemetic regimen prescribed along with chemotherapy and 3) to determine patient satisfaction with the calendar study tool.

ELIGIBILITY:
Inclusion criteria:

* Outpatients 18 years or older receiving chemotherapy treatment for neoadjuvant or adjuvant solid organ cancers,
* Able to provide consent for themselves,
* Calendar was only available in the English language, thus fluency in English was required.

Exclusion criteria:

* Participants who did not attain a minimum of grade 8 education,
* Significant visual impairment that precluded the ability to read the picture-based medication calendar,
* Difficulty swallowing with requirement for liquid formulations of medications,
* If planned to receive multiple cycles of chemotherapy at satellite oncology location instead of main study site,
* If unable to repeat the instructions back to research personnel or a care provider had to speak on the participant's behalf, the participant was withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Medication Adherence to Prescribed Antiemetics | 1 year
  Adherence is quantified as the number of doses taken of a prescribed agent divided by the number of doses prescribed, expressed as a percentage. Pill counts were utilized to calculate the number of missed doses or pills taken as a percentage of the total number prescribed and dispensed.

SECONDARY OUTCOMES:
Patient Understanding and Satisfaction Survey | 1 year
  The participant survey conducted at end of study was investigator-created and asked questions regarding demographics and medication taking behaviors. Questions specifically related to the calendar for those in the intervention arm were also asked. Questions regarding satisfaction with the calendar as well as complexity of medication regimen for oncologic treatment were assessed using a 5-point Likert scale.
Medication Use and Self-Efficacy (MUSE) Scale | 1 year
  19 The tool measures an individual's perceived ability to understand information about prescribed medicines, and to follow instructions for use.

CONTACTS AND LOCATIONS:
Overall Officials: Venita Harris, PharmD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No